CLINICAL TRIAL: NCT07072221
Title: A Prospective, Exploratory Clinical Study of Bendamustine Combined With Chidamide and Lenalidomide for Relapsed and Refractory Peripheral T-cell Lymphoma Patients
Brief Title: Bendamustine Combined With Chidamide and Lenalidomide for Relapsed and Refractory PTCL Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024473
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Bendamustine; Chidamide; Lenalidomide
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (ASCT-eligible) (Experimental): Patients who achieved PR/CR after 6 cycles of BCL regimen and were eligible to ASCT will proceed to ASCT consolidation
  Interventions: Drug: BCL regimen; Procedure: Cohort 1 (ASCT-eligible)
- Cohort 2 (ASCT-ineligible) (Experimental): Patients who achieved PR/CR after 6 cycles of BCL regimen and were ineligible to ASCT will receive oral chidamide maintenance therapy (minimum 2 years or until progression/unacceptable toxicity)
  Interventions: Drug: BCL regimen; Drug: Cohort 2 (ASCT--ineligible)

INTERVENTIONS:
Drug: BCL regimen — Induction therapy period (28 days*6)
  Bendamustine; Specification: 100mg per vial; 90mg/m2 d1-2, ivgtt.; for age≤70 years; 70mg/m2 d1-2, ivgtt.; for age>70 years;
  Chidamide; Specification: 5mg per tablet; 20mg biw for 2 weeks, po.; for age≤70 years; 15mg biw for 2 weeks, po.; for age>70 years;
  Lenalidomide Specification:10mg per tablet; 10mg qd d1-d21, po.; for age≤70 years; 10mg qd d1-d14, po.; for age>70 years;
Procedure: Cohort 1 (ASCT-eligible) — Autologous hematopoietic stem cell transplantation
  SEAM conditioning
  Simustine 250mg/m2 orally, d1;
  Etoposide 200mg/m2 intravenous infusion, d2-d5;
  Cytarabine 400mg/m2 intravenous infusion, d2-d5;
  Metformin 140mg/m2 intravenous infusion, d6;
  Arms: Cohort 1 (ASCT-eligible)
Drug: Cohort 2 (ASCT--ineligible) — Maintenance therapy period (2 years)
  Chidamide; Specification: 5mg per tablet; 15mg biw for 2 weeks per 3 weeks, po.;
  Arms: Cohort 2 (ASCT-ineligible)

SUMMARY:
To evaluate the efficacy and safety of bendamustine combined with chidamide and lenalidomide in R/R PTCL patients.

DETAILED DESCRIPTION:
This study will enroll relapsed/refractory (R/R) peripheral T-cell lymphoma (PTCL) patients aged over 18 years who have received at least one line of prior systemic therapy. Participants will receive combination therapy with bendamustine, chidamide, and lenalidomide (BCL regimen), with dose reduction for patients >70 years old. After 4 cycles of BCL regimen, patients demonstrating stable disease(SD) or progressive disease (PD) will be withdrawn from the study. Patients achieving partial remission(PR) or complete remission(CR) will receive another 2 cycles of BCL regimen followed by stratification treatment as followings:

Cohort 1 (ASCT-eligible): Responders will proceed to autologous stem cell transplantation (ASCT) consolidation

Cohort 2 (ASCT-ineligible): Responders will receive oral chidamide maintenance therapy (minimum 2 years or until progression/unacceptable toxicity)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female not limited;
2. Patients must have the capacity to understand and willingly provide written informed consent;
3. ECOG score 0-3 points;
4. Expected lifespan>3 months;
5. Patients with peripheral T-cell lymphoma (PTCL) confirmed by histopathology/cytology using the 2022 World Health Organization (WHO) Classification of Diseases;
6. Measurable lesions with a short diameter of ≥15mm defined by PET/CT;
7. R/R PTCL: patients with at least previous first-line treatment failure and no prior exposure to chidamide, lenalidomide and bendamustine;
8. Any non-hematological toxicity, except hair loss, associated with prior treatment in patients with R/R disease, as per NCI CTCAE version 5.0, must be managed and resolved to at least grade 1;
9. Appropriate organ function: Cardiac function: ejection fraction ≥ 50%, asymptomatic arrhythmia; Liver function: alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal, total bilirubin<2 times the upper limit of normal; Renal function: serum creatinine clearance rate ≥ 80 mL/min, creatinine<160 umol/l; Pulmonary function: Without oxygen inhalation, SPO2>90%, FEV1, FVC, and DLCO ≥ 50% predicted values;
10. Adequate bone marrow reserve is defined as: Hemoglobin ≥ 9g/dL, Platelet count ≥ 70 × 10 ^ 9/L, The absolute value of neutrophils is ≥ 1.0 × 10 ^ 9/L, If accompanied by bone marrow invasion, platelet count ≥ 50 × 10 ^ 9/L, absolute neutrophil count ≥ 0.75 × 10 ^ 9/L, The number of CD34+cells is ≥ 2.0 × 109/kg;
11. Subjects with fertility or potential for fertility must be willing to undergo contraception from the date of registration in this study until the study follow-up period;
12. Patients with good compliance.

Exclusion Criteria:

1. Patients with R/R disease previously used chidamide, lenalidomide and bendamustine, or received any other anti-tumor therapy within 4 weeks.
2. Patients enrolled in another clinical study within 4 weeks;
3. HIV infection and/or active hepatitis B or C;
4. Uncontrolled active infections;
5. Severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine>3 times the upper limit of normal);
6. Existence of organic heart disease or severe arrhythmia, leading to clinical symptoms or abnormal heart function (NYHA functional class ≥ 2);
7. Simultaneously present other tumors that require treatment or intervention;
8. Previous or current history of vascular embolism;
9. Pregnant or lactating women;
10. In a state of severe immune suppression;
11. Other psychological conditions that hinder patients from participating in research or signing informed consent forms.
12. Patients are unlikely to complete all protocol study visits and procedures or do not meet the requirements for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate(CRR) | At the end of 4 cycles of BCL regimen (each cycle is 28 days)
  The rate of patients who achieved CR after 4 cycles of bendamustine combined with chidamide and lenalidomide therapy (BCL regimen).

SECONDARY OUTCOMES:
Main adverse events | From enrollment to 1 month after the end of last patient's treatment
  The safety and tolerability of the BCL regimen measured by the major adverse events.
Overall response rate(ORR) | At the end of 4 cycles of BCL regimen (each cycle is 28 days)
  The rate of patients who achieved CR or PR after treatment of 4 cycles of BCL regimen
2-year Overall survival(OS) | From enrollment to 2 years after the last patient's treatment
  OS will be assessed from the start of the BCL treatment to the date of death or end of follow-up.
2-year progression-free survival(PFS) | From enrollment to 2 years after the last patient's treatment
  PFS will be assessed from the start of the BCL treatment to the date of progression, relapse, death or end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No